CLINICAL TRIAL: NCT05606380
Title: A Phase I Clinical Study to Investigate the Safety, Tolerability and Pharmacokinetic Characteristics of HLX60 (Anti-GARP Monoclonal Antibody) in Subjects With Advanced/Metastatic Solid Tumors or Lymphoma
Brief Title: A Phase I Study to Investigate the Safety, Tolerability and PK of HLX60 (Anti-GARP Monoclonal Antibody) in Subjects With Solid Tumors or Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX60-102
Record Dates: First submitted 2022-11-01; First posted 2022-11-04 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2023-08

CONDITIONS: Solid Tumor and Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HLX60 Group (Experimental): The initial dose of HLX60 is 0.5mg/kg, and 5 dose levels are designed: 2mg/kg, 5mg/kg, 15mg/kg and 25mg/kg (Q3W). Patients will receive the treatment until without any clinical benefit, death, intolerable toxicity, or withdraw the informed consent (whichever occurs first)
  Interventions: Drug: HLX60

INTERVENTIONS:
Drug: HLX60 — HLX60(anti-GARP Monoclonal Antibody）have 5 dose cohorts: 0.5, 2, 5, 15, 25mg/kg, intravenous infusion, every 3 weeks.

SUMMARY:
This trial is an open, dose escalation phase I clinical study. Subjects can only enter this study after they meet the inclusion and exclusion criteria.Into subjects will accept HLX60 intravenous infusion, every 3 weeks, treatment until lose clinical benefit, toxicity, death, revocation of informed consent.

ELIGIBILITY:
Key Inclusion Criteria:

1. Aged ≥ 18, ≤75 years at the time of signing the ICF;
2. Patients with histologically or cytologically confirmed advanced malignant solid tumor or lymphoma, who have failed or cannot receive the standard treatment;
3. With at least one evaluable lesion according to RECIST V1.1 (for solid tumors) or the Lugano criteria (for lymphomas);
4. Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 1 at enrollment;
5. Expected survival > 3 months;
6. Have appropriate organ functions;
7. The first administration of the investigational product must be: at least 28 days apart from the previous major surgery, medical device treatment, or local radiotherapy; at least 21 days apart from the previous cytotoxic chemotherapy, immunotherapy, and biological agent therapy; at least 14 days apart from the previous hormone therapy and surgical operation; at least 21 days or 5 half-lives apart from the administration of small molecule targeted drugs, whichever is longer; at least 14 days apart from the traditional Chinese medicine for tumor indications;
8. For patients with hepatocellular carcinoma, Child-Pugh score has to be A;
9. Male and female subjects with child-bearing potential must agree to use at least one highly effective contraception method during the study and within at least 6 months after the last administration of the investigational product.

Key Exclusion Criteria:

1. Have had other malignant tumors within 3 years before enrollment, except: (a) those with cured cervical carcinoma in situ or non-melanoma skin cancer; (b) those with cured second primary cancer without recurrence within 3 years; (c) those with double primary cancers believed to be able to benefit from this study; (d) those whose metastasis has been clearly excluded from a certain primary tumor source;
2. A history of (non-infectious) interstitial lung disease (ILD) requiring steroid use, current ILD, or a suspicion of ILD cannot be ruled out by imaging at screening; Note: Patients with radiation pneumonitis judged to be mild by the investigator can be enrolled.
3. The adverse reactions (except alopecia and other adverse reactions determined by the investigator to have no safety risk) of previous anti-tumor therapy have not yet recovered to ≤ grade 1 (CTCAE V5.0);
4. Those who are known to have severe anaphylaxis (grade 4 or greater in CTCAE V5.0) to macromolecular protein preparations/monoclonal antibodies or to any component of the investigational product;
5. Patients with any of the following unstable or poorly controlled diseases:1)Active systemic infectious diseases requiring intravenous antibiotics within 2 weeks before the first administration of the investigational product;2)Any poorly-controlled cardiovascular and cerebrovascular clinical symptoms or diseases, including but not limited (1) NYHA Class II or greater cardiac failure or left ventricular ejection fraction (LVEF) <50%;（2）unstable angina pectoris； (3) myocardial infarction and cerebral infarction within 6 months, (4) clinically significant supraventricular or ventricular arrhythmia without clinical intervention or poorly controlled after clinical intervention;3)Other chronic diseases which, in the opinion of the investigator, may compromise the safety of the patient or the integrity of the study;
6. Assessed as unsuitable for inclusion by the investigator, due to brain metastases, spinal cord compression, or cancerous meningitis with clinical symptoms, or uncontrolled brain or spinal cord metastases that have been evidenced; Note: Patients with asymptomatic or stable brain metastases, spinal cord compression, or carcinomatous meningitis as judged by the investigator were eligible for enrollment.
7. Those who have received anti-GARP or anti-GARP/TGF-β antibody therapy;
8. Have active autoimmune diseases (including but not limited to the following diseases or syndromes, such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism), except: vitiligo or cured childhood asthma/allergy that does not need any intervention in adulthood, autoimmune mediated hypothyroidism treated with stable dose of thyroid replacement hormone, and type I diabetes treated with stable dose of insulin; those in a stable condition and requiring no systemic immunosuppressant therapy (including corticosteroid hormone) are allowed to be enrolled;
9. Have received systemic corticosteroids (prednisone > 10 mg/d or equivalent dose of similar drug) or other immunosuppressants within 14 days before the first administration; Except: patients treated with topical, ocular, intra-articular, intranasal, and inhaled corticosteroids; those with short term use of corticosteroids for prophylaxis, such as contrast agents;
10. Patients in pregnancy [confirmed by serum beta-human chorionic gonadotropin (ß-HCG) test] or breastfeeding;
11. With a history of immunodeficiency, including human immunodeficiency virus (HIV)-positive or other acquired or congenital immunodeficiencies, or a history of organ transplantation;
12. Have active tuberculosis。
13. Active HBV, HCV infection or co-infection;
14. Have received live vaccines within 28 days prior to the first administration;
15. Patients whose medical history or any other evidence suggests that participation in the study may confuse the results, or subjects for whom the investigator believes the study is not in their best interest.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
DLT | from day1 to day 21
  The Dose-Limiting Toxicity (DLT) of HLX60 within 3 weeks after the first Administration in patients with Advanced/Metastatic Solid Tumors or Lymphomas
MTD | from day1 to day 21
  The Maximum Tolerated Dose (MTD) of HLX60 within 3 weeks after the first Administration in patients with Advanced/Metastatic Solid Tumors or Lymphomas

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, College of medicine, Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No